CLINICAL TRIAL: NCT04369729
Title: A Multidisciplinary Translational Approach to Investigate the Mechanisms, Predictors, and Prevention of Persistent Post-Traumatic Headache - Human Studies Protocol: Individual Projects Excluding Clinical Trial
Brief Title: Investigate the Mechanisms, Predictors, and Prevention of Persistent Post-Traumatic Headache
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Arizona (Other); Translational Genomics Research Institute (Other); Arizona State University (Other); Phoenix VA Health Care System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Amgen (Industry)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Other Study IDs: 20-003732
Record Dates: First submitted 2020-04-25; First posted 2020-04-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Post-Traumatic Headache: Individuals who have post-traumatic headache attributed to mild traumatic brain injury according to ICHD-3 diagnostic criteria
- Healthy Control: Healthy controls will have no history of traumatic brain injury and no history of migraine or other headaches

SUMMARY:
This is a United States Department of Defense funded Focused Program study that aims to identify mechanisms and predictors for persistent of post-traumatic headache attributed to mild traumatic brain injury, and identify methods of preventing post-traumatic headache persistence

DETAILED DESCRIPTION:
The human studies component of this Focused Program include clinical phenotyping, neurophysiology, molecular and genetic biomarker discovery, and brain imaging. This data will be utilized to characterize post-traumatic headache and build univariate and multivariate predictive models for post-traumatic headache persistence and for the response to post-traumatic headache treatment. Some participants might be eligible to participate in the clinical trial portion of this study.The clinical trial is a double-blind, randomized, placebo-controlled investigation of erenumab for the treatment of post-traumatic headache. Participants will be randomized when PTH has been present for 35-56 days. The clinical trial component of this Focused Program is described in more detail in a separate clinicaltrials.gov record.

Follow-up questionnaires, headache diary data, pain threshold results, and brain imaging data will be collected longitudinally during the trial to assess for changes over time and associations of such changes with post-traumatic headache treatment outcomes.

ELIGIBILITY:
POST-TRAUMATIC HEADACHE ELIGIBILITY CRITERIA

Inclusion Criteria:

* Have a diagnosis of acute PTH attributed to mild traumatic injury to the head as defined by the International Classification of Headache Disorders (ICHD-3).
* PTH onset 7-56 days prior to the time of enrollment.
* Adults 18-70 years of age.
* Willing to maintain a headache diary.
* Willing and able to return for follow-up visits.

Exclusion Criteria:

* Chronic headache (i.e. at least 15 headache days/month for more than 3 months) within 12 months prior to the mTBI that led to the current PTH, including PPTH, chronic migraine, medication overuse headache, new daily persistent headache, hemicrania continua, chronic tension-type headache.
* Diminished decision-making capacity that in the investigator's opinion would interfere with the person's ability to provide informed consent and complete study procedures.
* Started or changed dose of a headache preventive medication within the 3 months prior to screening.
* Use of onabotulinumtoxinA in the head, neck or face region within 6 months of screening.
* During the 6 months before screening, use of opioids or barbiturates on at least 4 days per month.
* Subjects who underwent an intervention or used a device (e.g., nerve blocks, transcranial magnetic stimulation, vagal nerve stimulation, or electrical trigeminal nerve stimulation) for headache.
* History of major psychiatric disorder such as schizophrenia and bipolar disorder.
* History or evidence of any unstable or clinically significant medical condition, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* History of positive neuroimaging findings that indicate a moderate or severe TBI.
* Contraindications to magnetic resonance imaging, including, but not limited to (only for those individuals participating in the MRI portion of this research):

  1. Metal implants
  2. Aneurysm clips
  3. Severe claustrophobia
  4. Implanted electronic devices
  5. Insulin or infusion pump
  6. Cochlear/otologic/ear implant
  7. Non-removable prosthesis
  8. Implanted shunts/catheters
  9. Certain intrauterine devices
  10. Tattooed makeup
  11. Body piercings that cannot be removed
  12. Metal fragments
  13. Wire sutures or metal staples
* Factors that reduce MR image quality and interpretability (only for those individuals participating in the MRI portion of this research):

  1. Dental braces or other non-removable devices (e.g., retainers)
  2. Prior brain surgery
  3. Known brain MRI abnormality that in the investigator's opinion will significantly impact MRI data.
* Sensory disorders that in the investigator's opinion might affect perception of cutaneous thermal stimuli (e.g., peripheral neuropathy) (only for those individuals undergoing pain threshold testing).
* Pregnancy
* Breastfeeding
* Currently or within 90 days prior to screening: received treatment in another drug study or an investigational device study.

HEALTHY CONTROL ELIGIBILITY CRITERIA

Inclusion Criteria:

* Adults 18-70 years of age.
* Willing and able to return for follow-up visits.

Exclusion Criteria:

* History of traumatic brain injury.
* History of migraine or other headaches (Tension-type headache up to an average of 3 days per month is allowed).
* Diminished decision-making capacity that in the investigator's opinion would interfere with the person's ability to provide informed consent and complete study procedures.
* During the 6 months before screening, use of opioids or barbiturates on an average of at least 4 days per month.
* History of major psychiatric disorder such as schizophrenia and bipolar disorder.
* History or evidence of any unstable or clinically significant medical condition, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Contraindications to magnetic resonance imaging, including, but not limited to:

  1. Metal implants
  2. Aneurysm clips
  3. Severe claustrophobia
  4. Implanted electronic devices
  5. Insulin or infusion pump
  6. Cochlear/otologic/ear implant
  7. Non-removable prosthesis
  8. Implanted shunts/catheters
  9. Certain intrauterine devices
  10. Tattooed makeup
  11. Body piercings that cannot be removed
  12. Metal fragments
  13. Wire sutures or metal staples
* Factors that reduce MR image quality and interpretability:

  1. Dental braces or other non-removable devices (e.g., retainers)
  2. Prior brain surgery
  3. Known brain MRI abnormality that in the investigator's opinion will significantly impact MRI data.
* Sensory disorders that in the investigator's opinion might affect perception of cutaneous thermal stimuli (e.g., peripheral neuropathy).
* Pregnancy
* Breastfeeding
* Currently or within 90 days prior to screening: received treatment in another drug study or an investigational device study
* Has previously received any CGRP ligand or receptor targeted monoclonal antibody

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be enrolled from the Mayo Clinic and Phoenix VA Healthcare System and from the surrounding region
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Longitudinal Assessment of PTH Phenotype | baseline with longitudinal follow-up at weeks four and sixteen
  descriptive analysis of post-traumatic headache characteristics such as headache frequency and severity, and characteristics of associated conditions such as symptoms of sensory hypersensitivities, anxiety, depression, insomnia, autonomic dysfunction, and cognitive function
Longitudinal Assessment of Cutaneous Pain Thresholds | baseline with longitudinal follow-up at weeks four and sixteen
  heat pain thresholds on the skin determined by quantitative sensory testing
Longitudinal Assessment of Visual Pain Thresholds from Bright Light Exposure | baseline with longitudinal follow-up at weeks four and sixteen
  visual pain thresholds to different light intensities
Longitudinal Assessment of Brain MRI | baseline with longitudinal follow-up at weeks four and sixteen
  structural brain imaging to include measures such as cortical thickness, regional volumes, brain curvature, white matter tract integrity, and functional brain imaging measures such as resting state functional connectivity and pain-induced brain activation
Longitudinal Assessment of Blood Based Biomarkers | baseline with longitudinal follow-up at weeks four and sixteen
  blood-based biomarkers, including DNA and targeted serum proteins, associated with acute and persistent post-traumatic headache and response to therapy
Longitudinal Assessment of Post-traumatic Headache Biomarkers | baseline with longitudinal follow-up at weeks four and sixteen
  clinical characteristics, pain thresholds, and brain imaging features as described above that are associated with acute post-traumatic headache and persistent post-traumatic headache; that predict the persistent of post-traumatic headache; and that predict and measure treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schwedt, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials